CLINICAL TRIAL: NCT00385762
Title: Effect of Selective Serotonin Reuptake Inhibitor Antidepressants on Semen Parameters
Brief Title: SSRI Effects on Semen Parameters in Men
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0605008515
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Human volunteers
MeSH Terms: interventions — Paroxetine; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples Semen samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: paroxetine — paroxetine 10-40mg daily x 5 weeks
  Other Names: Selective Serotonin Reuptake Inhibitor (SSRI)

SUMMARY:
According to the National Institute of Mental Health, depressive disorders afflict over six million U.S. men annually. Most cases of moderate or severe depression are treated with antidepressants, including monoamine oxidase inhibitors, tricyclic antidepressants, and, more recently, selective serotonin reuptake inhibitors (SSRIs) and antidepressants with modest serotonin and norepinephrine reuptake inhibition but unknown mechanism-of-action. Over the past two years, prescribing data show a steady increase in antidepressant dispensing rates (especially including serotonin reuptake inhibitors) for adults. SSRIs are known to have an effect on ejaculatory function and are therapeutically used for treatment of premature (rapid) ejaculation. However, few studies have evaluated the potential impact of antidepressant medications on male fertility, and no studies have been published with respect to the impact of newer antidepressants, such as SSRIs, on male fertility. In the high-volume male infertility practice at New York Hospital-Cornell Medical Center, several patients have presented who have had a clear temporal association between SSRI use and impairment in sperm motility and/or sperm transport (emission). These men have shown improvement in sperm counts and motility after discontinuation of antidepressant medications.

DETAILED DESCRIPTION:
We propose a crossover pilot study of normal healthy males to ascertain possible effects of SSRIs on semen parameters. After initial screening semen analyses, subjects will take the SSRI paroxetine for five weeks. Serial semen analyses will be obtained while on medication and one month after discontinuation of medication. Comparisons between semen parameters on and off medication will be used to evaluate the frequency and significance of semen analysis changes during SSRI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy male volunteers, ages 18-65
* Must be able to swallow pills

Exclusion Criteria:

* Known sexual dysfunction
* Tobacco use
* Prescription medications
* History of psychiatric disorders
* Previous chemotherapy or radiation treatment
* History of seizure disorder
* Alcohol use greater than 2 ounces daily
* Illicit drug use
* Azoospermia on screening semen analysis
* Varicocele
* Currently attempting to achieve pregnancy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter N. Schlegel, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Department of Urology, Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Paroxetine: Paroxetine was administered for 5 weeks using an escalating dosing schedule: week 1, 10 mg daily; week 2, 20 mg daily; weeks 3 and 4, 30 mg daily; week 5, 20 mg daily.
Period: Overall Study
Arm/Group | Paroxetine
Started | 35
Completed | 33
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paroxetine
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Semen Volume
Description: measured in mL
Time Frame: 2 months post initial visit
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Paroxetine
Number analyzed (Participants) | 33
mL | 2.55 (1.26)

2. Primary Outcome: Sperm Concentration
Description: number of sperm per cubic centimeter of semen
Time Frame: 2 months post initial visit
Measure: Mean (Standard Deviation); unit: number of sperm per cubic centimeter
Arm/Group | Paroxetine
Number analyzed (Participants) | 33
number of sperm per cubic centimeter | 75 (67.65)

3. Primary Outcome: Sperm Motility
Description: percent of sperm with movement
Time Frame: 2 months post initial visit
Measure: Mean (Standard Deviation); unit: Percent of sperm with movement
Arm/Group | Paroxetine
Number analyzed (Participants) | 33
Percent of sperm with movement | 50.21 (16.55)

4. Primary Outcome: Sperm Morphology
Description: percent of sperm with normal shape
Time Frame: 2 months post initial visit
Measure: Mean (Standard Deviation); unit: percent of sperm with normal shape
Arm/Group | Paroxetine
Number analyzed (Participants) | 33
percent of sperm with normal shape | 20.24 (8.89)

ADVERSE EVENTS:
Arm/Group | Paroxetine
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paroxetine (N=33)
Side effect to medication (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes